CLINICAL TRIAL: NCT03657680
Title: Description of Joint Range of Motion, Muscular Strength and Functionality of Patients Submitted to Total Hip Arthroplasty.
Brief Title: Range of Motion, Muscular Strength and Functionality of Patients Submitted to Total Hip Arthroplasty.
Status: Completed | Type: Observational
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Bruna de Moraes Lopes, Prof, Federal University of Health Science of Porto Alegre
Other Study IDs: THA patients evaluation
Record Dates: First submitted 2018-08-15; First posted 2018-09-05 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ATQ Group: Convenience sample of patients from Porto Alegre (RS, Brazil) who were experiencing unilateral hip osteoarthritis and were submitted to THA in referral hospitals at least five months previously to data collection. The volunteers were submitted to an evaluation of pain, range of motion, muscular strength and functional capacity.
  Interventions: Other: Evaluation
- Control Group: The control group was composed of asymptomatic individuals from the community. The volunteers were submitted to an evaluation of pain, range of motion, muscular strength and functional capacity.
  Interventions: Other: Evaluation

INTERVENTIONS:
Other: Evaluation — The volunteers were submitted to an evaluation of pain, range of motion, muscular strength and functional capacity.

SUMMARY:
Subjects in the late postoperative phase (5-8 months) of THA and control subjects without any signs or symptoms in the hip joint will be assessed for functionality (Harris Hip Score questionnaire and Timed Up and Go test), level of pain (visual analogue pain scale), hip range of motion and muscle isometric peak torque. This evaluation will be performed in order to compare functionality, level of pain, hip range of motion and peak torque between patients following total hip arthroplasty (THA) and asymptomatic controls.

DETAILED DESCRIPTION:
A descriptive, comparative cross-sectional study will be conducted. Participants will attended the Physical Therapy Laboratory at the Federal University of Health Sciences of Porto Alegre in a single assessment session. This study was approved by the university's Research Ethics Committee (protocol 925.402) and, prior to data collection, all participants will read and sign a consent form.

The experimental group will be composed of a convenience sample of patients from Porto Alegre (RS, Brazil) who were experiencing unilateral hip osteoarthritis and were submitted to THA in referral hospitals at least five months previously to data collection. Medical record information will be obtained from computerized hospital systems and potential participants will be invited by telephone to take part in the study. The control group will be composed of asymptomatic individuals from the community.

Participants will be considered eligible for the study if: they are at least 50 years old; have not undergone previous surgery and/or injection of corticosteroids to lower limb joints; have no clinical signs of osteoarthritis in other lower limbs joints; and experienced no disabling neurological or cardiovascular conditions. Individuals who have developed complications (infections, deep vein thrombosis and/or dislocation of the prosthetic component) during the postoperative period will be excluded.

Level of hip pain will be assessed using a 10-cm visual analog scale. It will be assessed in two stages: before (pre) and after completion of data collection (post-evaluation). Functional capacity will be assessed using the Timed Up and Go test and the Harris Hip Score questionnaire. To perform the Timed Up and Go test, subjects will be instructed to stand up from an armless chair and walk 3m, at their usual speed, to a mark drawn on the floor, then turn around, return to the chair and sit. The test will firstly be demonstrated by the evaluator and then performed by the participant twice, however only the second performance will be timed. Harris Hip Score is a hip joint assessment instrument; its score ranges from 0 to 100 points, consisting of pain, function, deformity and range of motion domains. The Harris Hip Score results will be classified according to the score, where: lower than 70 points is bad; between 70-79 is normal; between 80-89 is good; and, between 90-100 is excellent. Active range of motion measures will be performed in both hips by a single examiner using a fleximeter (FL6010 model, Sanny, Brazil). The protocol is adapted from the instrument manual, so that movements are assessed in the following positions: hip flexion, lying in supine and with knee flexed; hip extension, abduction and adduction, in standing position; and hip internal and external rotation, with the patient sitting on the edge of the table, with hip and knee flexed at 90º [21]. Movements will be interrupted if the second evaluator observes any compensation at the pelvis and/or trunk. The order of evaluation (affected or unaffected limb first) for fleximetry and dynamometry will be randomized using a mobile application (Randomizers - www.random.org). Hip muscles will be assessed isometrically using a BiodexTM Multi Joint System 4 Pro isokinetic dynamometer (Biodex Medical Systems, New York, USA). Equipment calibration will be performed according to the instructions in the manufacturer's manual. The chair is going to be set with 0° of inclination and the greater trochanter will be used as reference for alignment of the lower limb rotation axis. Participants' position is going to be maintained using stabilizing braces around the trunk, pelvis and contralateral limb. Patients position will took into account the postoperative limitations of THA and will be based on previous literature. Both hip flexors and extensors will be evaluated with the patient in a supine position, the tested limb in 45° of hip flexion and the contralateral limb in extension (image 1). Resistance platform will be set ~3cm above the upper limit of the patella. Both hip abductors and adductors assessments are going to be performed in side lying (image 2), the tested limb placed in 15° of hip abduction with the resistance platform lateral to the thigh, as the contralateral limb remained in flexion. Each muscle group evaluation will be preceded by an explanation of the test, as well as submaximal muscle contractions for familiarization and warm-up. Three attempts of 5s duration will be performed for each muscle group, with a 90s interval between each. Participants will be stimulated to exert their maximum strength during each attempt through verbal encouragement by the examiner.

ELIGIBILITY:
Inclusion Criteria:

* Age equal or superior to 50 years;
* have undergone a surgical procedure of unilateral total hip arthroplasty (cemented, non-cemented and hybrid prostheses) for at least 5 months and at most 18 months;
* referred by orthopedic physicians in the city of Porto Alegre or whose information (date of surgery, telephone contact, age and sex) were obtained through access to the computerized system in the physiotherapy sector of reference hospitals;
* who read and consent to the Informed Consent Form and understood the orientations necessary for the evaluation proposed in this study.

Exclusion Criteria:

* Performing a surgical procedure on other joints in the lower limbs;
* previous surgical procedures in the hip joint; osteoarticular diseases in lower limb joints;
* presence of signs or symptoms of contralateral hip osteoarthrosis;
* performed intra-articular injection of corticosteroids in the lower limbs during the last six months;
* cardiovascular diseases with the presence of disability, such as severe dyspnea and uncontrolled arterial hypertension;
* history of labyrinthitis;
* diabetes mellitus with signs of peripheral neuropathy and the presence of neurological diseases.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients submited to unilateral total hip arthroplasty and healthy subjects, with no signs and symptons envolving hip joint.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Isometric Muscle Strenght - Biodex | 1 hour
  Hip muscle isometric strenght were assessed isometrically using a BiodexTM Multi Joint System 4 Pro isokinetic dynamometer (Biodex Medical Systems, New York, USA). Flexor, extensor, abductor and adductor muscle strength were measured.

SECONDARY OUTCOMES:
Functionality - Timed Up and Go | 2 minutes
  Evaluation of patients functionality according to the performance in the Timed Up and Go Test. Subjects were instructed to stand up from an armless chair and walk 3m, at their usual speed, to a mark drawn on the floor, then turn around, return to the chair and sit. The test will be firstly demonstrated by the evaluator and then performed by the participant twice, however only the second performance will be timed.
Functionality - Harris Hip Score | 10 minutes
  Harris Hip Score is a hip joint assessment instrument; its score ranges from 0 to 100 points, consisting of pain, function, deformity and range of motion domains. The Harris Hip Score results were classified according to the score, where: lower than 70 points was bad; between 70-79 was normal; between 80-89 was good; and, between 90-100 was excellent. The scale evaluates pain, functionality, gait and mobility.
Joint Range of Motion | 20 minutes
  Active range of motion measures were performed in both hips by a single examiner using a phleximeter (FL6010 model, Sanny, Brazil). The protocol was adapted from the instrument manual, so that movements were assessed in the following positions: hip flexion, lying in supine and with knee flexed; hip extension, abduction and adduction, in standing position; and hip internal and external rotation, with the patient sitting on the edge of the table, with hip and knee flexed at 90º [21]. Movements were interrupted if the second evaluator observed any compensation at the pelvis and/or trunk.
Pain Intensity Evaluation | 5 minutes
  Pain in the hip joint was evaluated with a 10cm Visual Analogue Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Bruna M Lopes, Prof, Principal Investigator — Federal University of Health Science of Porto Alegre

IPD SHARING:
Plan to Share IPD: No